CLINICAL TRIAL: NCT00617799
Title: Pilot Study to Identify Biomarkers That May Predict Response to High Dose IL-2
Brief Title: Biomarkers That Predict Response to High-Dose Aldesleukin in Metastatic Kidney Cancer or Metastatic Melanoma
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0278-07-FB; P30CA036727 (NIH)
Record Dates: First submitted 2008-02-15; First posted 2008-02-18 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: stage IV renal cell cancer; stage IV melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — aldesleukin; Gene Expression Profiling; Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected prior to, at mid-course and at the end of the course of IL-2 therapy.

INTERVENTIONS:
Biological: aldesleukin
Genetic: gene expression analysis
Genetic: mutation analysis
Other: flow cytometry

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at biomarkers that predict response to high-dose aldesleukin in patients with metastatic kidney cancer or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship of peripheral blood lymphocyte phenotype pattern in patients with metastatic renal cell carcinoma or metastatic melanoma to response to high-dose aldesleukin (IL-2).
* Determine the relationship of peripheral blood mononuclear cells gene microarray patterns in patients with metastatic renal cell carcinoma or metastatic melanoma to response to high-dose IL-2.
* Determine the frequency of mutations on genes encoding for IL-2 receptor A and B.

OUTLINE: Patients receive high-dose aldesleukin (IL-2) as part of standard treatment on days 1 and 8. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline, prior to beginning course 2, and 4 weeks after the completion of course 2. Samples are analyzed using peripheral blood cytometry, gene microarray analysis, and IL-2 receptor single-nucleotide polymorphism techniques.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic renal cell carcinoma or metastatic melanoma
* Must be receiving treatment with high-dose aldesleukin as part of standard therapy

Exclusion Criteria:

none

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be receiving HD IL-2.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-10-02 (Actual); Primary Completion 2009-02-18 (Actual); Study Completion 2010-04-16 (Actual)

PRIMARY OUTCOMES:
Relationship of peripheral blood lymphocyte phenotype to response to high-dose aldesleukin (IL-2) | 10 weeks
  Relationship of peripheral blood lymphocyte phenotype to response to high-dose aldesleukin (IL-2) from blood draws at baseline, prior to course 2 and 4 weeks after course 2
Relationship of peripheral blood mononuclear cells gene microarray patterns to response to high-dose IL-2 | 10 weeks
  Relationship of peripheral blood mononuclear cells gene microarray patterns to response to high-dose IL-2 from blood draws at baseline, prior to course 2 and 4 weeks after course 2
Frequency of mutations on genes encoding IL-2 receptor A and B | 10 weeks
  Frequency of mutations on genes encoding IL-2 receptor A and B from blood draws at baseline, prior to course 2 and 4 weeks after course 2

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hauke, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Eppley Cancer Center, Omaha, Nebraska, United States